CLINICAL TRIAL: NCT06587256
Title: Mouth Tape for Snoring and Sleep Apnea (MTASSA)
Brief Title: Study to Examine the Effect of Silicone Mouth Tape on Snoring and Mild Sleep Apnea.
Acronym: MTASSA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00425791
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Mild Obstructive Sleep Apnea; Snoring
Keywords: sleep apnea; snoring; mouth tape
MeSH Terms: conditions — Snoring; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label, non-randomized interventional clinical trial comparing each participant's baseline snoring or sleep apnea level to the participant's 3-month snoring or sleep apnea while using mouth tape during sleep.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simple snorers or Mild Sleep Apnea (Experimental): Patients with snoring and a prior sleep study showing an AHI < 15.
  Interventions: Device: Mouth Tape

INTERVENTIONS:
Device: Mouth Tape — A single piece of silicone tape placed vertically over the lips. When positioned properly the participant can still inhale/exhale and cough around the tape if needed, but will tend to keep mouth closed otherwise.

SUMMARY:
Snoring is a common problem caused by vibration of tissues in the throat region during sleep. Although snoring is sometimes dismissed as a minor nuisance rather than a medical disorder, several studies indicate that snoring can disrupt sleep quality of the snorer, as well as the snorer's bed partner. Snoring also might lead to problems such as dry mouth, bad breath, dental problems, and even cardiovascular disease. Current treatments for snoring include lifestyle modifications such as weight loss, side-sleeping, and avoidance of evening alcohol intake. In some cases, invasive surgeries, dental devices, or even CPAP are recommended for snoring. These interventions have mixed effectiveness and may be difficult to use.

It may be possible to treat snoring by fostering nasal breathing, while avoiding mouth-breathing during sleep. Breathing through the mouth reduces the airway diameter and contributes to snoring. Several studies show that nasal breathing can reduce snoring volume and improve airflow. Recent studies have shown that covering the mouth during sleep with adhesive patches or tape can improve snoring volume without adverse effects. However, these studies were performed in a small number of patients and did not fully measure the impact of the intervention on sleep quality, sleep architecture, or the experience of the bed partner, who is often the overlooked "victim" of the snoring. In this interventional study, the investigators will examine the safety and efficacy of mouth tape for snoring, focusing on subjective and objective snoring/breathing metrics of both the snorer and bed partner.

Snoring is sometimes also a sign of obstructive sleep apnea (OSA). If OSA is ruled out with a sleep study, patients are considered to have "simple" snoring. When OSA is mild (apnea hypopnea index 15), treatments can include the same interventions as snoring (e.g. weight loss, avoidance of alcohol, side-sleeping) or can be more aggressively treated with devices such as continuous positive airway pressure (CPAP). CPAP may be challenging to use, expensive, and associated with side effects such as mouth dryness and skin irritation. Alternative, inexpensive, and well-tolerated interventions are needed for mild OSA. For this reason, the investigators include patients with snoring and mild OSA in this study.

DETAILED DESCRIPTION:
Snoring affects hundreds of millions of people worldwide and describes vibration of airway tissues including the palate, tongue, tonsils, and epiglottis. In a random sample of middle-aged adults, habitual snoring was reported by 45%. Snoring decreases the sleep quality of the snoring individual and the snorer's bed partner, causes social stigma, and may lead bed partners to sleep in separate rooms. Snoring may also be a manifestation of obstructive sleep apnea (OSA), in which the upper airway collapses partially or fully, leading to episodic pauses in breathing (apneas) or shallow breathing (hypopneas). While many physicians and patients recognize health risks of OSA, snoring is often dismissed as "benign" or "simple", but this is a misnomer. Heavy snoring per se can contribute to unrefreshing sleep and daytime fatigue. In study of 400 adult women who underwent polysomnography, snoring was associated with daytime sleepiness, even after adjustment for the presence of OSA. Data from a home sleep apnea testing device equipped with a snoring microphone found that loud sustained snoring predicted daytime sleepiness better than intermittent bursts of sound characteristic of OSA. Other studies suggest that snoring may increase risks of carotid atherosclerosis which could increase the chances of a stroke. A study of surgery for simple snoring reported improvements in marital life after surgery illustrating the impact of snoring and its resolution on sleep quality and relational health. Hence, snoring is a highly prevalent problem that impairs the sleep quality of snorers and the snorer's bed partner.

Current approaches to snoring include weight loss, avoidance of tobacco and alcohol, lateral sleep, nasal decongestants or steroids, nasal dilator adhesive devices, surgeries, or devices (such as CPAP or mandibular advancement devices). Most of these therapies are recommended on the basis of anecdotes and small studies. Insurance generally does not cover CPAP or oral appliances for simple snoring. Despite the nearly ubiquitous nature of snoring, there is no well-researched standard of care.

A large proportion of air enters and exits the nose during typical awake breathing. During sleep some people breathe more orally, which predisposes to snoring and OSA by increasing upper airway resistance and decreasing retro-glossal and retro-palatal area. Under sedation, mouth opening caused a significant increase in the upper airway critical pressure indicating a greater likelihood of airway obstruction compared to mouth closure. Using an oronasal ("full face") mask with a partition installed between the nose and mouth, closure of the nasal port caused severe OSA, which resolved after closing only the mouth port to force nasal breathing, or opening both ports to allow spontaneous breathing. CPAP applied via an oronasal mask is less effective than CPAP applied via a nasal mask. In recent studies, mouth occlusion with a plastic barrier device or silicone tape dramatically reduced snoring volume, and lowered the apnea hypopnea index (AHI) in patients with mild OSA or simple snoring. Mouth closure with a barrier device also improved the performance of an oral appliance for treatment of OSA. These studies demonstrate that mouth breathing predisposes to snoring and OSA, and that diverting breathing through the nose can reduce snoring. However, these studies are limited by small sample size, a homogenous population (Asian men with normal BMI), short study duration, and lack of input from the bed partner.

This project investigates the efficacy of mouth tape in two common clinical scenarios. First, the scenario of a patient with simple snoring after OSA has been ruled out. These patients are typically prescribed lifestyle modification (weight loss, avoidance of supine sleep, tobacco and alcohol) or non-prescription remedies such as nasal dilator strips or decongestant sprays. The second scenario is a patient presenting with snoring and few other symptoms who is found to have mild OSA (apnea hypopnea index, AHI 15). While the treatment for mildly symptomatic mild OSA is debated, the first line therapy is typically CPAP or lifestyle modification. Adherence to CPAP is notoriously challenging. Even among patients who use CPAP chronically, there are frequent side effects such as skin abrasions. Mouth tape might be another treatment option for these patients.

The investigators justify the combined inclusion of snoring patients and those with mild OSA in this study for several reasons. First, overlap in physiology: the same individual may be diagnosed with simple snoring on one night and mild OSA on another, as snoring and OSA are caused by inspiratory flow limitation, which may manifest as night-to-night variability of AHI on sleep studies. Second, overlap in evidence-based management: patients with mild OSA are often managed similarly to simple snorers, since the necessity of CPAP (or other therapies) for mild OSA is controversial. Third, overlap in clinical need: there is significant demand for alternative effective and well-tolerated treatments for both conditions.

In the clinical setting of simple snoring or mild OSA, the investigators will offer patients the option of mouth tape during sleep. A small piece of silicone mouth tape is placed vertically over the lips without fully occluding the mouth, which the investigators hypothesize will lower snoring volume and improve sleep quality for the snorer and bed partner. Patients will be carefully screened who tolerate nasal breathing and have no other complicating cardiopulmonary disease. In consented patients the investigators will measure the safety and tolerability of mouth tape, and the impact of mouth tape on sleep and snoring as perceived by the patient and bed partner after 3 months.

Interestingly, mouth taping has become a viral social media trend with the hashtag mouth taping (#mouthtaping) on Tiktok reaching 160 million views as of 1/5/2024. Many of these posts make bold claims about improved sleep quality, improved sinuses, and even lower blood pressure with mouth taping. The medical community has been slow and uncertain in its response to this phenomenon, illustrating the need for more rigorous research.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a body mass index of 35 kg/m2 with a self-reported history of snoring and a bed partner who can provider answers to about the patients snoring. Patients must have a prior sleep study that shows no sleep apnea, or mild sleep apnea (AHI under 15 events/hr).

Exclusion Criteria:

* Allergy to silicone mouth tape, chronic lung disease, facial hair preventing wearing of the tape
* Grade 3+ or 4+ tonsils, prior palatal or tongue surgery.
* Patients may not have any form of chronic or acute hypoventilation.
* Patients must be able to tolerate breathing through their nose with the mouth tape in place for at least 3 minutes.
* Patients may not be pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Snoring / Sleep Survey (SSS) | Baseline and 3 months
  The patient will be asked about perceived snoring and sleep quality (score range 0-25, best=0, worst =25)

SECONDARY OUTCOMES:
Adherence and tolerance questionnaire | 3 months
  Asks about ease of use and any intolerances (score range 0-100, hard = 0, 100=easy).
Sleep apnea severity (WatchPAT) | Baseline and 3 months
  The investigators will use a home sleep apnea test. Sleep apnea severity will be scored based on peripheral arterial tonometry (PAT)-signal derived apnea hypopnea index (pAHI).
Snoring intensity (WatchPAT) | Baseline and 3 months
  The investigators will use a home sleep apnea test. Snoring intensity be me measured using vibration assessment to derive estimate decibels (dB).
PROMIS Sleep Related Disturbance (SD) Short Form 8A (PROMIS-SD-8A) | Baseline, 2 weeks, and 3 months
  PROMIS-SD 8a questionnaire asks about perceived sleep quality (score range 0 - 40, 0=very poor, 40=very good)
PROMIS Sleep Related Impairment (SRI) Short Form 8A (PROMIS-SRI-8A) | 2 weeks
  PROMIS-SRI 8a questionnaire asks about sleep and its impact on daytime function (score range 0 - 40, 0=very impaired, 40=not at all impaired)
Snoring / Sleep Survey (SSS) Bed Partner | Baseline, 2 weeks, and 3 months
  The bed partner will be asked about the participants snoring, and the bed partner's own sleep quality (score range 0-25, best=0, worst =25).
Snoring / Sleep Survey (SSS) Patient | 2 weeks
  The patient will be asked about snoring and sleep quality (score range 0-25, best=0, worst =25).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Jun, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
If requested, a de-identified data set including only participant age, sex, weight, height, questionnaire, and sleep study data will be provided.
Supporting Information: Study Protocol
Time Frame: The individual participant data (IPD) will be available at the termination of the study and accessible for 2 years after study closure.
Access Criteria: Requests must be provided to the P.I. in writing with documentation supporting the need for access. If appropriate a de-identified data set will be provided via an encrypted file.

REFERENCES:
- [Background] Lee YC, Lu CT, Cheng WN, Li HY. The Impact of Mouth-Taping in Mouth-Breathers with Mild Obstructive Sleep Apnea: A Preliminary Study. Healthcare (Basel). 2022 Sep 13;10(9):1755. doi: 10.3390/healthcare10091755. PMID 36141367
- [Background] Huang TW, Young TH. Novel porous oral patches for patients with mild obstructive sleep apnea and mouth breathing: a pilot study. Otolaryngol Head Neck Surg. 2015 Feb;152(2):369-73. doi: 10.1177/0194599814559383. Epub 2014 Dec 1. PMID 25450408